CLINICAL TRIAL: NCT06935838
Title: Effects of Tirzepatide on Weight Loss and Chronic Inflammation in People With HIV
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Hawaii (Other)
Responsible Party: Principal Investigator, Christine Akamine, Assistant Professor, University of Hawaii
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H064
Record Dates: First submitted 2025-04-04; First posted 2025-04-20 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Obesity and Overweight; HIV; Chronic Inflammation
MeSH Terms: conditions — Obesity; Overweight | interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tirzepatide (Experimental)
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — Tirzepatide is approved by the Food and Drug Administration (FDA) for the treatment of type 2 diabetes, obesity and overweight with at least one weight-related medical condition, and moderate to severe obstructive sleep apnea. An initial dose of TZP 2.5 mg subcutaneous (SQ) once weekly will be given, escalated by 2.5 mg at 4-week intervals to a final dose of 7.5mg.

SUMMARY:
This is a prospective cohort study of 12 overweight (with one or more weight-related condition) or obese adults with well controlled HIV-1 on antiretroviral therapy (ART). An initial dose of tirzepatide (TZP) 2.5 mg subcutaneous (SQ) once weekly will be given, escalated by 2.5 mg at 4-week intervals to a final dose of 7.5mg. The investigators will collect the following information via review of the medical record: age, race/ethnicity, sex, medical conditions, medications, most recent standard of care HIV labs (including T-cell panel and HIV-1 viral load). The primary outcome will be the change in baseline body weight at 12 weeks. Secondary outcomes will be changes in body composition, liver fat content and liver stiffness, inflammatory markers, cardiometabolic markers (lipids and HbA1c), and monocytes at 12 weeks. There will be a 4-week safety follow up off TZP.

ELIGIBILITY:
Age ≥ 18 years

HIV-1 infection (well controlled)

* Documented HIV-1 infection ≥ 1 year prior to study entry (ELISA confirmed by Western blot or HIV-1 RNA) AND
* HIV-1 RNA <200 copies/mL for ≥ 6 months

Stable ART

· Receiving a stable antiretroviral regimen for at least 1 year prior to study entry

Overweight

* BMI ≥27 kg/m2 plus at least one weight-related condition (defined as a medical history of dyslipidemia, hypertension, cardiovascular disease, or obstructive sleep apnea) OR Obese
* BMI ≥ 30 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Baseline Body Weight | 12 weeks
  The primary outcome will be the change in baseline body weight (measured in lbs) at 12 weeks.

SECONDARY OUTCOMES:
Change in Inflammatory Markers: GM-CSF | 12 weeks
  All biomarkers will be assayed from banked plasma using a Luminex multiplex assay and ELISAs performed per manufacturer's instructions. A Cytokine 10-Plex Human Panel (ThermoFisher Scientific) with data acquired using Luminex 200TM system (Luminex) and ELISAs (ThermoFisher Scientific) with data acquired using a Victor X3 plate reader (PerkinElmer) will be utilized to measure the following inflammatory biomarkers: GM-CSF. Cytokine standards supplied by the manufacturer will be run in duplicate on each plate.
Change in cardiometabolic markers | 12 weeks
  We will evaluate HbA1c and a lipid profile at the baseline, week 12 and week 16 study visits.
Monocyte Subset Analysis | Week 12 and week 16
  Monocyte subsets will be phenotyped from thawed/washed banked cryopreserved PBMCs (from blood drawn at baseline, week 12, and week 16) using a multiparametric panel of conjugated monoclonal antibodies: CD3, CD14, CD16, CD56, CD19, CD20, HLA-DR antibodies with Live/Dead fixable yellow dead cell stain (YARD). Data will be acquired on a 4-laser BD LSRFortessa Flow Cytometer with all compensation and gating analyses performed with the FlowJo analytical software to determine levels of classical (CD14 ++ CD16 -), intermediate (CD14 ++ CD16 +), non-classical (CD14 + CD16 ++), and transitional (CD14 + CD16 -) monocytes.
Change in Inflammatory Markers: IFN-γ | 12 weeks
  All biomarkers will be assayed from banked plasma using a Luminex multiplex assay and ELISAs performed per manufacturer's instructions. A Cytokine 10-Plex Human Panel (ThermoFisher Scientific) with data acquired using Luminex 200TM system (Luminex) and ELISAs (ThermoFisher Scientific) with data acquired using a Victor X3 plate reader (PerkinElmer) will be utilized to measure the following inflammatory biomarkers: IFN-γ. Cytokine standards supplied by the manufacturer will be run in duplicate on each plate.
Change in Inflammatory Markers: IL-1β | 12 weeks
  All biomarkers will be assayed from banked plasma using a Luminex multiplex assay and ELISAs performed per manufacturer's instructions. A Cytokine 10-Plex Human Panel (ThermoFisher Scientific) with data acquired using Luminex 200TM system (Luminex) and ELISAs (ThermoFisher Scientific) with data acquired using a Victor X3 plate reader (PerkinElmer) will be utilized to measure the following inflammatory biomarkers: IL-1β. Cytokine standards supplied by the manufacturer will be run in duplicate on each plate.
Change in Inflammatory Markers: IL-2 | 12 weeks
  All biomarkers will be assayed from banked plasma using a Luminex multiplex assay and ELISAs performed per manufacturer's instructions. A Cytokine 10-Plex Human Panel (ThermoFisher Scientific) with data acquired using Luminex 200TM system (Luminex) and ELISAs (ThermoFisher Scientific) with data acquired using a Victor X3 plate reader (PerkinElmer) will be utilized to measure the following inflammatory biomarkers: IL-2. Cytokine standards supplied by the manufacturer will be run in duplicate on each plate.
Change in Inflammatory Markers: IL-1β, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10 | 12 weeks
  All biomarkers will be assayed from banked plasma using a Luminex multiplex assay and ELISAs performed per manufacturer's instructions. A Cytokine 10-Plex Human Panel (ThermoFisher Scientific) with data acquired using Luminex 200TM system (Luminex) and ELISAs (ThermoFisher Scientific) with data acquired using a Victor X3 plate reader (PerkinElmer) will be utilized to measure the following inflammatory biomarkers: IL-1β, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10. Cytokine standards supplied by the manufacturer will be run in duplicate on each plate.
Change in Inflammatory Markers: TNF-α | 12 weeks
  All biomarkers will be assayed from banked plasma using a Luminex multiplex assay and ELISAs performed per manufacturer's instructions. A Cytokine 10-Plex Human Panel (ThermoFisher Scientific) with data acquired using Luminex 200TM system (Luminex) and ELISAs (ThermoFisher Scientific) with data acquired using a Victor X3 plate reader (PerkinElmer) will be utilized to measure the following inflammatory biomarkers: TNF-α. Cytokine standards supplied by the manufacturer will be run in duplicate on each plate.
Change in Inflammatory Markers: NFkB | 12 weeks
  All biomarkers will be assayed from banked plasma using a Luminex multiplex assay and ELISAs performed per manufacturer's instructions. A Cytokine 10-Plex Human Panel (ThermoFisher Scientific) with data acquired using Luminex 200TM system (Luminex) and ELISAs (ThermoFisher Scientific) with data acquired using a Victor X3 plate reader (PerkinElmer) will be utilized to measure the following inflammatory biomarkers: NFkB. Cytokine standards supplied by the manufacturer will be run in duplicate on each plate.
Change in Inflammatory Markers: sCD163, and sCD14 | 12 weeks
  All biomarkers will be assayed from banked plasma using a Luminex multiplex assay and ELISAs performed per manufacturer's instructions. A Cytokine 10-Plex Human Panel (ThermoFisher Scientific) with data acquired using Luminex 200TM system (Luminex) and ELISAs (ThermoFisher Scientific) with data acquired using a Victor X3 plate reader (PerkinElmer) will be utilized to measure the following inflammatory biomarkers: sCD163, and sCD14. Cytokine standards supplied by the manufacturer will be run in duplicate on each plate.
Body composition | 12 weeks
  Body composition (total, peripheral and truncal fat, and lean tissue) by dual energy absorptiometry (DEXA)
Waist circumference | 12 weeks
  Changes in waist circumference over 12 weeks of therapy
Liver fat content | 12 weeks
  Changes in Liver fat content (Controlled Attenuation Parameter, CAP) over 12 weeks
Liver stiffness measurement (LSM) | 12 weeks
  Changes in Liver stiffness measurement (LSM) over 12 weeks

OTHER OUTCOMES:
Biorepository samples for future research | The biorepository samples (only) will be banked for future analysis for separate research (related or unrelated to this project) for up to 7 years post-study completion.
  Obtaining blood specimens for banking in the biorepository for future analyses (frozen for retrospective analysis) related to HIV, cardiometabolic diseases, inflammation and the immune system. Biorespository specimens will be collected at baseline, week 12, week 16 and early discontinuation visits. It will not include genetic testing. The biorepository will enable the development of new hypotheses to further contribute toward understanding of HIV, the immune system, chronic inflammation, and cardiometabolic disease.

CONTACTS AND LOCATIONS:
Locations (1):
- John A Burns School of Medicine, Honolulu, Hawaii, United States

REFERENCES:
- [Background] Morisako AK, Tauali'i M, Ambrose AJH, Withy K. Beyond the Ability to Pay: The Health Status of Native Hawaiians and Other Pacific Islanders in Relationship to Health Insurance. Hawaii J Med Public Health. 2017 Mar;76(3 Suppl 1):36-41. PMID 28435757
- [Background] Hoagland A, Kipping S. Challenges in Promoting Health Equity and Reducing Disparities in Access Across New and Established Technologies. Can J Cardiol. 2024 Jun;40(6):1154-1167. doi: 10.1016/j.cjca.2024.02.014. Epub 2024 Feb 28. PMID 38417572
- [Background] Liang H, Xie Z, Shen T. Monocyte activation and cardiovascular disease in HIV infection. Cell Mol Immunol. 2017 Dec;14(12):960-962. doi: 10.1038/cmi.2017.109. Epub 2017 Oct 30. No abstract available. PMID 29082920
- [Background] Apovian CM, Aronne LJ, Bessesen DH, McDonnell ME, Murad MH, Pagotto U, Ryan DH, Still CD; Endocrine Society. Pharmacological management of obesity: an endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2015 Feb;100(2):342-62. doi: 10.1210/jc.2014-3415. Epub 2015 Jan 15. PMID 25590212
- [Background] Wharton S, Lau DCW, Vallis M, Sharma AM, Biertho L, Campbell-Scherer D, Adamo K, Alberga A, Bell R, Boule N, Boyling E, Brown J, Calam B, Clarke C, Crowshoe L, Divalentino D, Forhan M, Freedhoff Y, Gagner M, Glazer S, Grand C, Green M, Hahn M, Hawa R, Henderson R, Hong D, Hung P, Janssen I, Jacklin K, Johnson-Stoklossa C, Kemp A, Kirk S, Kuk J, Langlois MF, Lear S, McInnes A, Macklin D, Naji L, Manjoo P, Morin MP, Nerenberg K, Patton I, Pedersen S, Pereira L, Piccinini-Vallis H, Poddar M, Poirier P, Prud'homme D, Salas XR, Rueda-Clausen C, Russell-Mayhew S, Shiau J, Sherifali D, Sievenpiper J, Sockalingam S, Taylor V, Toth E, Twells L, Tytus R, Walji S, Walker L, Wicklum S. Obesity in adults: a clinical practice guideline. CMAJ. 2020 Aug 4;192(31):E875-E891. doi: 10.1503/cmaj.191707. No abstract available. PMID 32753461
- [Background] Jastreboff AM, Aronne LJ, Ahmad NN, Wharton S, Connery L, Alves B, Kiyosue A, Zhang S, Liu B, Bunck MC, Stefanski A; SURMOUNT-1 Investigators. Tirzepatide Once Weekly for the Treatment of Obesity. N Engl J Med. 2022 Jul 21;387(3):205-216. doi: 10.1056/NEJMoa2206038. Epub 2022 Jun 4. PMID 35658024
- [Background] Nguyen Q, Wooten D, Lee D, Moreno M, Promer K, Rajagopal A, Tan M, Tang M, Duren K, Yin J, Hill L. Glucagon-like Peptide 1 Receptor Agonists Promote Weight Loss Among People With HIV. Clin Infect Dis. 2024 Oct 15;79(4):978-982. doi: 10.1093/cid/ciae151. PMID 38501237
- [Background] Crum-Cianflone N, Tejidor R, Medina S, Barahona I, Ganesan A. Obesity among patients with HIV: the latest epidemic. AIDS Patient Care STDS. 2008 Dec;22(12):925-30. doi: 10.1089/apc.2008.0082. PMID 19072098
- [Background] Lv T, Cao W, Li T. HIV-Related Immune Activation and Inflammation: Current Understanding and Strategies. J Immunol Res. 2021 Sep 29;2021:7316456. doi: 10.1155/2021/7316456. eCollection 2021. PMID 34631899
- [Background] Lenharo M. Obesity drugs have another superpower: taming inflammation. Nature. 2024 Feb;626(7998):246. doi: 10.1038/d41586-024-00118-4. No abstract available. PMID 38278941
- [Background] Todosenko N, Khaziakhmatova O, Malashchenko V, Yurova K, Bograya M, Beletskaya M, Vulf M, Mikhailova L, Minchenko A, Soroko I, Khlusov I, Litvinova L. Adipocyte- and Monocyte-Mediated Vicious Circle of Inflammation and Obesity (Review of Cellular and Molecular Mechanisms). Int J Mol Sci. 2023 Jul 31;24(15):12259. doi: 10.3390/ijms241512259. PMID 37569635
- [Background] Sotak M, Clark M, Suur BE, Borgeson E. Inflammation and resolution in obesity. Nat Rev Endocrinol. 2025 Jan;21(1):45-61. doi: 10.1038/s41574-024-01047-y. Epub 2024 Oct 24. PMID 39448830
- [Background] Yanovski SZ, Yanovski JA. Approach to Obesity Treatment in Primary Care: A Review. JAMA Intern Med. 2024 Jul 1;184(7):818-829. doi: 10.1001/jamainternmed.2023.8526. PMID 38466272